CLINICAL TRIAL: NCT03435289
Title: A Phase I Study of CPI-613 in Combination With Gemcitabine and Nab-paclitaxel (Abraxane) for Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: A Study of CPI-613 With Gemcitabine and Nab-paclitaxel for Patients With Advanced or Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Collaborators: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA CPI 613
Record Dates: First submitted 2017-11-17; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — devimistat; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label study of CPI-613 in combination with gemcitabine and nab-paclitaxel for patients with locally advanced or metastatic pancreatic cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613, Gemcitabine and Nab-paclitaxel (Other): CPI-613 in Combination With Gemcitabine 1000mg/m2 iv and Nab-paclitaxel 125mg/m2 iv
  Interventions: Drug: CPI 613 in Combination With Gemcitabine and Nab-paclitaxel

INTERVENTIONS:
Drug: CPI 613 in Combination With Gemcitabine and Nab-paclitaxel — Day 1,15 CPI-613: IV infusion at a rate of 4 mL/min via a central venous catheter starting at 500 mg/m2 (with concurrent D5W infusing at a rate of 125-150 cc/hr). The CPI dose will be determined based on cohort. Day 2,16 Neulasta as clinically indicated
  Nab- paclitaxel 125mg/m2 iv over 30 min followed by Gemcitabine 1000mg/m2 iv over 30 min
  Other Names: Gemcitabine; Nab-paclitaxel; Abraxane; Gemzar

SUMMARY:
This is a single arm, open-label study of CPI-613 in combination with gemcitabine and nab-paclitaxel for patients with locally advanced or metastatic pancreatic cancer never treated with systemic chemotherapy.

DETAILED DESCRIPTION:
The primary specific aim of the study is to establish the maximum tolerated dose (MTD) of CPI-613 when given in combination with gemcitabine/nab-paclitaxel for patients with locally advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented and measurable stage III or IV pancreatic adenocarcinoma.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. First line treatment for patients diagnosed with metastatic disease
4. First line treatment for patients with locally advanced pancreatic cancer who have not been treated with systemic therapies. Prior treatment with chemoradiation is allowed if 4 or more weeks have passed from completion of chemo-radiotherapy.
5. Expected survival > 3 months.
6. Women of child-bearing potential must use accepted contraceptive methods (abstinence, intrauterine device, oral contraceptive, or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
7. Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
8. Laboratory values ≤2 weeks must be:

   A. Adequate hematologic (platelet count ≥ 100,000 cells/mm^3 or ≥ 100 bil/L; absolute neutrophil count [ANC] ≥ 1500 cells/mm3 or ≥1.5 bil/L; and hemoglobin ≥ 9 g/dL or ≥ 90 g/L).

   B. Adequate hepatic function (aspartate aminotransferase [AST/SGOT] ≤ 3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] ≤ 3x UNL (≤ 5x UNL if liver metastases present), Total bilirubin ≤ 1.5x ULN C. Adequate renal function (serum creatinine ≤ 2.0 mg/dL or 177 μmol/L). D. Adequate coagulation (International Normalized Ratio or INR must be ≤ 1.5), unless the patient receives anticoagulation treatment in which case the INR should be within the therapeutic level, not higher than 3.5 E. Albumin > 2.5 g/dL
9. No evidence of active infection and no serious infection within the past month.
10. Mentally competent, ability to understand and willingness to sign the informed consent form.

    -

Exclusion Criteria:

1. Unwilling or unable to follow protocol requirements. Endocrine or acinar pancreatic carcinoma
2. Known cerebral metastases, central nervous system (CNS), or epidural tumor
3. Prior treatment with any systemic chemotherapy for metastatic adenocarcinoma of the pancreas or for stage III (locally advanced) adenocarcinoma
4. Presence of clinically significant abdominal ascites
5. Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 2 weeks prior to initiation of CPI-613 treatment.
6. Serious medical illness that would potentially increase patients' risk for toxicity.
7. Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease).
8. Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown).
9. Lactating females.
10. Fertile men unwilling to practice contraceptive methods during the study period.
11. Life expectancy less than 3 months.
12. Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.
13. Unwilling or unable to follow protocol requirements.
14. Active heart disease including but not limited to symptomatic congestive heart failure (NYHA class 3 or 4), symptomatic coronary artery disease, symptomatic angina pectoris, or symptomatic myocardial infarction.
15. Patients with a history of myocardial infarction that is <3 months prior to registration.
16. Evidence of active infection, or serious infection within the past month.
17. Patients with known HIV infection.
18. Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of CPI-613 treatment. Steroid use for contrast induced allergy or other supportive care indication is allowed
19. Requirement for immediate palliative treatment of any kind including surgery.
20. Any other malignancy within last 3 years
21. History of interstitial lung disease, idiopathic pulmonary fibrosis or pulmonary hypersensitivity pneumonitis
22. Peripheral neuropathy grades 2 or higher

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The maximally tolerated dose of CPI 613 combined with Gemcitabine and nab-paclitaxel | Evaluation at monthly intervals through study completion from the date of study entry until the date of progression, up to 1 year

SECONDARY OUTCOMES:
The number of participants with treatment related adverse events as assessed by CTCAE v 4.0 | Evaluation at 2 week intervals through study completion from the date of study entry until the date of progression, up to 1 year
The number of participants with complete or partial response | Evaluation at 2 month intervals through study completion from the date of study entry until the date of progression, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Angela T Alistar, MD, Principal Investigator — Morristown Medical Center
Locations (2):
- United States (2):
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Medical Center, Summit, New Jersey

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available to other researchers